CLINICAL TRIAL: NCT00453518
Title: Evaluating the Use of the FiberNet® Embolic Protection System in Saphenous Vein Grafts: The RETRIEVE Study
Brief Title: The RETRIEVE Study: Use of the FiberNet® Embolic Protection System in Saphenous Vein Grafts
Acronym: RETRIEVE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Lumen Biomedical (Industry)
Responsible Party: Jill Moland, Sr. CRA, Lumen Biomedical, Inc.
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 90-1004
Record Dates: First submitted 2007-03-28; First posted 2007-03-29 (Estimated); Last update posted 2009-08-18 (Estimated); Status verified 2009-08

CONDITIONS: Saphenous Vein Graft Disease; Myocardial Ischemia; Embolism
Keywords: SVG; Saphenous Vein Graft; Embolic Protection; Distal Protection; EPD; FiberNet; Saphenous Vein Graft intervention
MeSH Terms: conditions — Myocardial Ischemia; Embolism | interventions — Stents

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Device: FiberNet EPS used during SVG intervention. — The FiberNet EPS is indicated for use as a guide wire and embolic protection system to capture and remove embolic material produced while performing percutaneous transluminal interventional procedures in saphenous vein grafts.
  Other Names: stenting

SUMMARY:
This is a multicenter, prospective study designed to demonstrate the performance and safety of the FiberNet Embolic Protection System when used as an adjunctive device during saphenous vein graft (SVG) intervention.

DETAILED DESCRIPTION:
The study will involve up to 30 patients to be enrolled using the FiberNet device during clinically indicated percutaneous intervention of SVG and followed through 30 days post procedure. Patients will be enrolled at up to 10 Investigative Sites. The study is a prospective multi-center registry with sequential enrollment of qualified patients who consent to participate and meet all entrance criteria.

The Lumen Biomedical, Inc. FiberNet® Embolic Protection System is indicated for use as a guide wire and embolic protection system to capture and remove embolic material (thrombus/debris) produced while performing percutaneous transluminal interventional procedures in saphenous vein grafts with reference vessel diameters of 1.75 mm to 7.0 mm.

ELIGIBILITY:
Inclusion Criteria:

* Candidate for percutaneous transluminal coronary angioplasty (PTCA), stenting and emergent coronary artery bypass graft (CABG).
* Myocardial ischemia as evidenced by one or more of the following:

  * Diagnosis of stable or unstable angina pectoris
  * ECG changes consistent with ischemia
  * Positive functional study
  * Recent myocardial infarction
* Lesion(s) is located within SVG and is ≥ 50% and < 100% stenosed.

Exclusion Criteria:

Clinical Criteria:

* Myocardial infarction with documented total CK-MB > 2 times the upper limit of normal within the past 24 hours, or currently experiencing an acute myocardial infarction.
* Undergone cardiac surgery within the past 60 days.
* A planned invasive surgical procedure within 30 days.
* The lesion(s) is in an SVG that is less than 2 months post-implant.
* Left ventricular ejection fraction < 20%.
* A stroke or transient ischemic neurological attack (TIA) within the past 2 months.

Angiographic Criteria:

* The lesion(s) is in an arterial conduit.
* Lesion is within 10 mm of the proximal anastomosis.
* More than two native lesions [in addition to the SVG lesion(s)] that need to be treated at the index procedure.
* More than two SVGs that need to be treated at the index procedure.
* Chronic total occlusion of a target lesion.
* The SVG lesion(s) requires treatment with a large device other than PTCA prior to stent placement (such as, but not limited to, directional coronary atherectomy, excimer laser, rotational atherectomy, rheolytic thrombectomy or brachytherapy).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2007-03; Primary Completion 2009-02 (Actual); Study Completion 2009-02 (Actual)

PRIMARY OUTCOMES:
The primary objective of the study is to evaluate the safety and performance of the FiberNet Embolic Protection System. The primary endpoint is major adverse cardiac events (MACE) rate at 30 days. | 30 days

SECONDARY OUTCOMES:
The secondary study objectives are endpoints related to the use of the FiberNet system and additional safety endpoints. | index hospitalization

CONTACTS AND LOCATIONS:
Overall Officials: Robert Feldman, MD — Munroe Regional Medical Center
Locations (6):
- United States (6):
  - Munroe Regional Medical Center, Ocala, Florida
  - St. Vincent Hospital, Indianapolis, Indiana
  - William Beaumont Hospital, Royal Oak, Michigan
  - Christ Hospital, Cincinnati, Ohio
  - Riverside Methodist Hospital, Columbus, Ohio
  - Lehigh Valley Hospital, Allentown, Pennsylvania

REFERENCES:
- See also: Lumen Biomedical website — http://www.lumenbio.com